CLINICAL TRIAL: NCT04351217
Title: Comparison Between the Use of Music and Relaxation Training on Craving Alcohol in Patients With Alcohol Dependence Syndrome: A Pilot Study
Brief Title: Music vs Relaxation Training in Craving Reduction in Alcohol Dependence Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasturba Medical College (Other)
Responsible Party: Principal Investigator, Shradha Chandrasekar, Student, MSc Clinical Psychology, Kasturba Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IEC KMC MLR 01-19/14
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Alcohol Dependence Syndrome
MeSH Terms: conditions — Alcoholism | interventions — Music Therapy; Autogenic Training

STUDY DESIGN:
Intervention Model Description: Two interventions, Music and Progressive Muscle Relaxation (PMR) were used. Music was Indian Classical Flute music, 23 minutes long. PMR was recorded for uniformity of delivery, and was 22 minutes in length.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Music was Indian Classical Flute music, 23 minutes long. It was played on a speaker at equal volume to ensure uniformity.
  Interventions: Behavioral: Music
- Progressive Muscle Relaxation (Experimental): Progressive Muscle Relaxation was recorded for uniformity of delivery, and was 22 minutes in length. It was played on a speaker at equal volume to ensure uniformity.
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Music — Raga Ahir Bhairav and Bhairavi were used, played primarily on flute, without lyrics.
  Arms: Music
Behavioral: Progressive Muscle Relaxation — The instructions were recorded in both English and the local language, Kannada
  Arms: Progressive Muscle Relaxation

SUMMARY:
The aim of the study was to compare the effectiveness of Music and Progressive Muscle Relaxation as interventions to reduce craving, increase coping, and understand the subjective experience of the interventions with patients diagnosed with Mental and Behavioral Disorders due to Alcohol, Dependence Syndrome, over a 5 day period.

DETAILED DESCRIPTION:
Craving for alcohol produces an aversive, uncomfortable state, with autonomic arousal similar to that in anxiety disorders, and is the main factor leading to relapse. Music has been shown to reduce anxiety and stress levels. Progressive Muscle Relaxation (PMR) is the intervention of choice for treatment of anxiety and related syndromes. This study aimed to compare efficacy of PMR and music in reducing levels of alcohol craving and increasing perceived ability to cope with the craving. The intervention was conducted over 5 days with two randomised group of 10 patients each. The patients were assigned to either group based on randomizer sequencing. Initial motivation was assessed before beginning the study. Measures of craving level and coping were collected on Day 1, 3 and 5. Single question exit interview was conducted to understand subjective perception of the patients regarding the techniques. Significant difference was found in coping levels through use of PMR (p = 0.01), and subjective reduction in craving levels was reported by patients in the music group, though this was not statistically significant. Thus, PMR may be used as an adjunct to increase coping abilities in patients with alcohol dependence, while music may be a useful tool to reduce craving but cannot be conclusively commented upon without further research.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Mental and Behavioral Disorders due to Use of Alcohol, Dependence Syndrome
* Abstinent for at least 1 week

Exclusion Criteria:

* Any other known psychiatric/physical condition
* Risk of Suicide or Relapse
* Less than 75% compliance

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Craving | 5 days
  The level of craving for alcohol experienced by the patient, as measured through Alcohol Urge Questionnaire.
Coping | 5 days
  The patient's perceived ability to cope with their craving for alcohol, as assessed through a visual analogue scale for coping

SECONDARY OUTCOMES:
Single Question Exit Interview | 5 days
  Each patient was a asked a single question during the final debriefing on the last day of the study. The question was "Please describe your experience with the music/exercise". Their answers were recorded verbatim and were translated from Kannada as needed

CONTACTS AND LOCATIONS:
Overall Officials: Keshava Pai Pai, MD, Study Chair — KMC Mangalore
Locations (1):
- KMC Mangalore, Mangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to confidentiality agreement.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT04351217/Prot_SAP_ICF_000.pdf